CLINICAL TRIAL: NCT00860964
Title: A Study of Prevention and Treatment of Postmenopausal Osteoporosis in Chinese Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMB 97-667
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Osteoporosis
Keywords: estradiol valerate; Medroxyprogesterone; menopause; Lipid; Bone mineral density; Body Composition
MeSH Terms: conditions — Osteoporosis | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- estradiol valerate (Experimental)
  Interventions: Drug: estradiol valerate

INTERVENTIONS:
Drug: Placebo — Placebo, calcium 900mg/d, VitD200iu/d and exercise
  Arms: Placebo
Drug: estradiol valerate — estradiol valerate 1mg/d,medroxyprogesterone 6mg/d for 10 days,calcium 900mg/d, VitD200iu/d and exercise
  Arms: estradiol valerate

SUMMARY:
The purpose of this trial is to study the efficacy and safety of low dose of estradiol valerate in the prevention and treatment of postmenopausal osteoporosis.

DETAILED DESCRIPTION:
Research purposes: To assess the Impact of hormone therapy on quality of life in early post-menopausal women; To assess the Impact of hormone therapy on cardiovascular system in early post-menopausal women; To assess the Impact of hormone therapy on cognitive function in early post-menopausal women; To assess the Impact of hormone therapy on osteoporosis in early post-menopausal women.

Study Design:

The clinical trial research was divided into 2 groups. Treatment group given estradiol valerate 1mg/d, periodic application of medroxyprogesterone 6mg/d for 10 days, calcium 900mg/d, VitD200iu/d and exercise(Brisk walking every day 2 times, continued for 10 minutes each time). Control group given placebo, calcium,VitD and exercise were same with treatment group.

ELIGIBILITY:
Inclusion Criteria:

All patients meet the criteria:

1. Patients with informed consent.
2. Breast Cancer inform possible danger.
3. Physical and mental health.

Menopausal transition meet the criteria:

1. Age between 40 ~ 55 years old.
2. Women with Menopause syndrome or menstrual disorders.
3. The second to fourth lumbar spine bone mineral density to normal.

Early postmenopause meet the criteria:

1. Age between 45 ~ 60 years old.
2. Spontaneous amenorrhea for more than six months and less than 5 years.
3. The second to fourth lumbar spine bone mineral density was between -1 and -2.5 Standard deviation Compared with normal young women.

Exclusion Criteria:

1. Tobacco or alcohol abuser.
2. History of various malignant diseases.
3. Women with Serious chronic diseases, such as liver and kidney dysfunction.
4. Women Suffering from endocrine diseases, such as Thyroid disease, Parathyroid disease,Adrenal disease and Osteomalacia.
5. Women with Long-term application of drugs, such as Antiepileptic drug, Adrenocorticotropic hormone, Diuretics and Heparin.
6. Women had used estrogen or calcitonin in the past 6 months.
7. Women has added higher than the physiological requirements VitD.
8. Who had taken bisphosphonates or sodium fluoride in the past 1 year.
9. Women had been taking Chinese medicines or other unregistered food in past 3 months.
10. Women with one of the following medical history or disease: Thrombophlebitis, estrogen-related thrombosis or thromboembolism, Cerebrovascular accident, with known or suspected estrogen-dependent tumor, undiagnosed vaginal bleeding, Cervical Pap smear graded at 3 or more, Serious uterine disorders, Serious breast disorders, Serious gallbladder disease, Severe hypertension and Hypercholesterolemia
11. Secondary osteoporosis.
12. Participants' lumbar spine anatomy(at least L1~L4) is not suitable to do dual-energy X-ray absorptiometry measured, such as obvious scoliosis, bone injury and Orthopedic surgery Sequelae.
13. Doctor consider inappropriate to participate in because of other diseases.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 1998-02; Primary Completion 2003-02 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 60 months

SECONDARY OUTCOMES:
ALT, Cr, TG, TC, HDL-C, LDL-C, Body Composition, Breast Ultrasound, Pelvic ultrasound | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Shou Q Lin, PhD, Principal Investigator — Gynecological endocrinology & women's health centre of Peking Union Medical College Hospital